CLINICAL TRIAL: NCT02515929
Title: Prospective Double-Blind Randomized Controlled Clinical Trial in the Gingivitis Prevention With an Oligomeric Proanthocyanidins Nutritional Supplement
Brief Title: Prospective Double-Blind Randomized Controlled Clinical Trial in the Gingivitis Prevention With OPCs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ROSA MARÍA DÍAZ SÁNCHEZ, DENTIST - MASTER STUDENT, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USeville
Record Dates: First submitted 2015-07-30; First posted 2015-08-05 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Gingivitis
Keywords: Oligomeric Proanthocyanidins; Periodontal Disease
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oligomeric Proanthocyanidins (Experimental): 90 mg exocian cran 408 plus 120mg Vitamin C, 1 tablet by mouth, every 24 hours for 21 days
  Interventions: Dietary Supplement: Oligomeric Proanthocyanidins
- Placebo (Placebo Comparator): Similar organoleptic experimental arm,1 tablet by mouth, every 24 hours for 21 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oligomeric Proanthocyanidins
  Arms: Oligomeric Proanthocyanidins
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Aim: To evaluate the effectiveness on tissue response of the new nutritional supplement made of Oligomeric Proanthocyanidins (OPCs) in induced gingivitis after 21 days of use.

Material and Methods: A double-blind randomized controlled prospective clinical trial was carried out on 20 patients divided into an experimental group treated with the OPCs pill and a control group treated with placebo, after fulfilling the selection criteria. Patients had to come 4 times during the study to register the Silness and Loe and Gingival Bleeding index, plaque index, inflammatory crevicular fluid study (IL6) and changes in brightness of the gingiva. No complementary hygiene methods were allowed during the 21 days.

DETAILED DESCRIPTION:
Material and Methods

Study Design and Population

A randomized, double-blind, placebo-controlled, clinical trial of 21 days of duration was conducted among 20 volunteer students of Dentistry of the University of Sevilla. No previous studies have been found in the literature, so 20 subjects were determined for the pilot study to test our hypothesis.

The study protocol was approved by the Ethics Committee of the University of Sevilla. Prior to participation, the purpose and procedures were fully explained to all patients and all participants gave written informed consent in accordance with Helsinki declaration. The study was designed, conducted, analysed and reported according to guidelines for Good Clinical Practice. The study was approved by the Clinical Trials.gov Protocol Registration and Results System with the number XXXXYY. The protocol can be accessed if necessary in ClinicalTrials.gov.

The study was carried out between September 2013 until January 2104. The recruitment started on September and the Baseline date took place on October 2013. After the 21 days follow-up, data was treated obtaining the results on January 2014.

At the pre-screening visit the Medical and Dental histories were taken and the screening was carried out base don the inclusion and exclusion criteria. Inclusion criteria were: subjects older than 18 years, male or female, good general health, a minimum of 20 teeth (teeth that have gross caries, were crowned or extensively restored, orthodontic banded, abutments, or third molars were not included in the tooth count), signed informed consent before study initiation.

Exclusion criteria were as follows: Periodontal disease, defined as 4 mm and / or positive bleeding on probing; Pregnant or breastfeeding; Subjects with fixed or removable prosthesis; Tumor pathology in oral cavity; Use of antibiotics during 2 months period prior to the start of the trial; Hypersensitivity to red fruits in general; Xerostomia; Active Smoker; Contagious-infectious pathologies; Pathology with severe systemic repercussions; Any other judgment of the investigator if he believes endangers or risk to the subject participant; Subjects with phenylketonuria or allergy to aspartame; Use of any oral hygiene product for the duration of the study.

A single examiner determined assessment of patient eligibility for the study and enrolment of patients into trial. Patients eligible for the study were individually randomly assigned to Oligomeric Proanthocyanidins Nutritional Supplement treatment or Placebo groups by an informatics programme by LACER S.A.

The study was double-blind. The examiner and the patient did not know into which group were assigned. Results were treated by another examiner who knows which patients belonged to the experimental or placebo group. The masking process was established by a number assignation to each patient in the study, the treatment was externally the same to the patient and examiner to not allowed knowing to which group belonged.

Patients had to take the experimental or placebo treatment each night after dinner and after rinse with water. The pill was maintained in the mouth until complete dissolution. Drink or eat was not allowed during 30 minutes after taking the treatment. The experimental treatment consisted on 90mg exocian cran 408 (equivalent to 36 mg OPC) and 120 mg of Vitamin C, while the placebo group was composed of the same organoleptic substance but free of active ingredients. Both were similar in appearance.

At the baseline stage of the trial a tartar removal was carried out in each patient and enough medication for the entire study plus a patient diary and instructions for its correct fulfilment were given. Inflammatory crevicular fluid (IL6) and the brightness of the gingiva were registered.

Two evaluation visits were performance on the day 14 and 21 after the baseline for an oral clinical examination and to register the Silness and Löe Index, the Gingival Bleeding index, the Turesky plaque index, inflammatory crevicular fluid study (IL6) and changes in brightness of the gingiva.

Silness and Löe index

Six teeth were examined according to Ramfjord criteria (16-21-24-36-41-44 ). Four surfaces of each tooth were examined, making a total of 24 measurements taken. These measurements were performance with a periodontal probe by the same examiner.

Gingival Bleeding index

A periodontal probe was used to make this index. The values established for the examination are found below:

0 - Absence of inflammation. 1 - Mild inflammation, slight change in colour and no gingival edema. No bleeding on probing. 2 - Moderate inflammation, redness, edema and gingival hypertrophy. Bleeds to probe (after 10 seconds). 3 - Severe inflammation, marked redness and hypertrophy. There may be ulcerations. Tends to spontaneous bleeding.

Turesky Plaque Index

The buccal surfaces of anterior teeth were examined using a mouthwash of basic fuchsine as developing agent plaque and a numerical scoring system from O to 5 was established.

0: There is no plaque 1: Independent streaks of plaque in the cervical margin of the tooth. 2: thin continuous band of plaque (up to 1mm) at the cervical margin. 3: Band greater than one millimetre wide, but covers less than one third of the crown. 4: The plate covers third but not more than two thirds of the crown. 5: The plate covers two thirds or more of the crown.

Inflammatory crevicular fluid study (IL6)

Crevicular fluid samples were collected from interdental areas (lingual, buccal, mesial, and distal) of six teeth distributed by the four quadrants (16, 21, 24, 36, 41 and 44) by 5 strips of pressed paper 2cm long, especially for crevicular fluid. The impregnation time for each patient was 5 seconds and immediately inserted into 0.5ml Eppendorf microtubes with 50ul saline at 4 ° C for preservation. The sample transport to the biological laboratory was in a refrigerator, being stored frozen at -80°C at the laboratory until being processed.

Then the investigator sproceeded to analyse the concentration (pg/ml) of interleukins 6 present in each sample using panels 96 well bioplex brand Luminex®.

Brightness of the Gingiva

The brightness of the gingiva was taken to identify possible changes in the gingival colour. The reddening of the gingiva accompanies the inflammation of the tissue, which is a factor that may help to differentiate inflammatory changes at this level.

The luminosity of the gingiva was registered with Micro SpectroShadeTM MHT Optic Research AG. This instrument is designed for taking dental colour. However, besides including colour guides, the SpectroShadeTM has the ability to measure the brightness of any colour, not just shades of white. The change in the colour of the gingiva was observed within the same patient measuring the reference colour for each patient in the same point in each evaluation visit and being able to compare the change in the coloration of the same point.

Statistical Data Treatment

The management of the data was performed using the SPSS statistical program. A similar database to Notebook Data Collection was created. For each variable a minimum and maximum range and the name of the variable and its values defined. The data are presented as the mean ± standard deviation of the measurements, and a p-value less than 0.05 was considered statistically significant.

Chi-square test was performed to qualitative variable, T-student to the quantitative variable, after the Kolmogorov Smirnov to assure the normality.

This study was approved by The Ethical Committee, and all examinations and treatments were performed with the consent of the subjects and according to the guidelines Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years, male or female, good general health, a minimum of 20 teeth (teeth that have gross caries, were crowned or extensively restored, orthodontic banded, abutments, or third molars were not included in the tooth count), signed informed consent before study initiation.

Exclusion Criteria:

* Periodontal disease, defined as 4 mm and / or positive bleeding on probing
* Pregnant or breastfeeding
* Subjects with fixed or removable prosthesis
* Tumor pathology in oral cavity; Use of antibiotics during 2 months period prior to the start of the trial; Hypersensitivity to red fruits in general; Xerostomia; Active Smoker; Contagious-infectious pathologies; Pathology with severe systemic repercussions; Any other judgment of the investigator if he believes endangers or risk to the subject participant; Subjects with phenylketonuria or allergy to aspartame; Use of any oral hygiene product for the duration of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Silness and Löe index | 21days
  Six teeth were examined according to Ramfjord criteria (16-21-24-36-41-44 ). Four surfaces of each tooth were examined, making a total of 24 measurements taken.
Gingival Bleeding index | 21 days
  A periodontal probe was used to make this index. The values established for the examination are found below:
  0 - Absence of inflammation. 1 - Mild inflammation, slight change in colour and no gingival edema. No bleeding on probing. 2 - Moderate inflammation, redness, edema and gingival hypertrophy. Bleeds to probe (after 10 seconds). 3 - Severe inflammation, marked redness and hypertrophy. There may be ulcerations. Tends to spontaneous bleeding.
Turesky Plaque Index | 21 days
  The buccal surfaces of anterior teeth were examined using a mouthwash of basic fuchsine as developing agent plaque and a numerical scoring system from O to 5 was established.
  0: There is no plaque 1: Independent streaks of plaque in the cervical margin of the tooth. 2: thin continuous band of plaque (up to 1mm) at the cervical margin. 3: Band greater than one millimetre wide, but covers less than one third of the crown. 4: The plate covers third but not more than two thirds of the crown. 5: The plate covers two thirds or more of the crown.
Inflammatory crevicular fluid study (IL6) | 21 days
  Crevicular fluid samples were collected from interdental areas (lingual, buccal, mesial, and distal) of six teeth distributed by the four quadrants (16, 21, 24, 36, 41 and 44) by 5 strips of pressed paper 2cm long, especially for crevicular fluid. The impregnation time for each patient was 5 seconds and immediately inserted into 0.5ml Eppendorf microtubes with 50ul saline at 4 ° C for preservation. The sample transport to the biological laboratory was in a refrigerator, being stored frozen at -80°C at the laboratory until being processed.
Brightness of the Gingiva | 21 days
  The brightness of the gingiva was taken to identify possible changes in the gingival colour. The reddening of the gingiva accompanies the inflammation of the tissue, which is a factor that may help to differentiate inflammatory changes at this level.
  The luminosity of the gingiva was registered with Micro SpectroShadeTM MHT Optic Research AG. This instrument is designed for taking dental colour. However, besides including colour guides, the SpectroShadeTM has the ability to measure the brightness of any colour, not just shades of white. The change in the colour of the gingiva was observed within the same patient measuring the reference colour for each patient in the same point in each evaluation visit and being able to compare the change in the coloration of the same point.